CLINICAL TRIAL: NCT01258660
Title: A Randomized, Double-blind, Double-dummy, 2-parallel Arms Clinical Trial to Assess the Pharmacodynamic Effect on Plasma Folate and Red Blood Cell Folate and to Compare the Profile of Circulating Folate Metabolites During 24 Weeks of Treatment With an Oral Contraceptive Containing Ethinylestradiol, Drospirenone and L-5-methyltetrahydrofolate (SH T04532A and SH T04532C) or Yasmin (SH T04532D and SH T04532PC) Co-administered With Folic Acid (SH K04532B) Followed by 20 Weeks of Open-label Treatment With Yasmin Only (Folate Elimination Phase) in Women Seeking Contraception
Brief Title: Assessment of the Pharmacodynamic Effect on Plasma Folate and Red Blood Cell Folate and Comparison of the Folate Metabolites During the 24 Weeks of Treatment (Yasmin + Metafolin Versus Yasmin + Folic Acid) Followed by a 20 Week Elimination Phase of Folate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 91509; 2006-003522-29 (EudraCT Number); 309763 (Other: Company Internal)
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Results first posted 2011-05-13 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Contraception
MeSH Terms: interventions — drospirenone; levomefolate calcium; drospirenone and ethinyl estradiol combination; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EE 0.03 mg/DRSP 3 mg/Metafolin + folic acid placebo (Experimental): Combination EE/DRSP/ Metafolin [0.030 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin] given orally in a cyclic regimen for 24 weeks (6 cycles) in combination with folic acid placebo tablets (encapsulated). Each treatment cycle consisting of once daily hormone and Metafolin treatment for 21-days followed by once daily hormone free, Metafolin only regimen for 7 days. This phase was followed by 20 weeks (5 cycles) folate elimination phase consisting of oral administration of Yasmin alone.
  Interventions: Drug: EE 0.03 mg/DRSP 3 mg/Metafolin + folic acid placebo
- EE 0.03 mg/DRSP 3 mg (Yasmin) + folic acid (Experimental): Yasmin [0.030 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP)] in combination with folic acid tablets 0.4 mg (encapsulated), given orally in a cyclic regimen for 24 weeks (6 cycles). Each treatment cycle providing once daily hormone and folic acid treatment for 21 days followed by once daily hormone free, folic acid only regimen for 7 days (encapsulated). This phase was followed by 20 weeks (5 cycles) folate elimination phase consisting of oral administration of Yasmin alone.
  Interventions: Drug: EE 0.03 mg/DRSP 3 mg (Yasmin) + folic acid

INTERVENTIONS:
Drug: EE 0.03 mg/DRSP 3 mg/Metafolin + folic acid placebo — Combination EE/DRSP/ Metafolin [0.030 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin] given orally in a cyclic regimen for 24 weeks (6 cycles) in combination with folic acid placebo tablets (encapsulated). Each treatment cycle consisting of once daily hormone and Metafolin treatment for 21-days followed by once daily hormone free, Metafolin only regimen for 7 days. This phase was followed by 20 weeks (5 cycles) folate elimination phase consisting of oral administration of Yasmin alone.
  Arms: EE 0.03 mg/DRSP 3 mg/Metafolin + folic acid placebo
Drug: EE 0.03 mg/DRSP 3 mg (Yasmin) + folic acid — Yasmin [0.030 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP)] in combination with folic acid tablets 0.4 mg (encapsulated), given orally in a cyclic regimen for 24 weeks (6 cycles). Each treatment cycle providing once daily hormone and folic acid treatment for 21 days followed by once daily hormone free, folic acid only regimen for 7 days (encapsulated). This phase was followed by 20 weeks (5 cycles) folate elimination phase consisting of oral administration of Yasmin alone.
  Arms: EE 0.03 mg/DRSP 3 mg (Yasmin) + folic acid

SUMMARY:
The purpose of this study is to examine and compare the uptake of levomefolate calcium (Metafolin, a registered vitamin supplement) and folic acid in the body during 24 weeks of treatment with a following folate elimination phase of 20 weeks in healthy volunteers seeking contraception. Yasmin (oral contraceptive containing drospirenone and ethinylestradiol) was co-administered over the entire period of 44 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years.
* RBC folate > 317 nmol/L and < 906 nmol/L.
* At least 1 menstruation during the last 3 months before screening with the exception of women using progestin-only methods (injection, implant) or progestin-releasing intrauterine system (IUS).
* Negative pregnancy test at screening and at admission into the study.
* Healthy as confirmed by medical history and physical examination.
* Body mass index (BMI) of 18.5-30.0 kg/m2 .
* Volunteers that smoke less than 10 cigarettes per day can be included up to the age of 30 years.
* Adequate vitamin B12 status defined as plasma B12 concentrations ≥ 110 pmol/L.

Exclusion Criteria:

* Regular intake of folic acid defined as > 100 μg folic acid/day in vitamin supplements or fortified food during the last 4 months.
* Treatment with the following medications, which has the potential of interfering with folate metabolism: cholestyramine, methotrexate, trimethoprim, sulfasalazine, salicylic acid, cotrimoxazol, antacids or antiepileptic drugs.
* Pregnancy, lactation (at least three cycles have to follow delivery, abortion, or lactation before start of treatment)
* Vascular or metabolic disease including existing or previous arterial thromboembolic diseases (myocardial infarction, stroke), existing or previous venous thromboembolic diseases (deep vein thrombosis, pulmonary embolism), and any condition which could increase the risk to suffer any of the above mentioned disorders
* Any disease or condition that could compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study medication.
* Any disease that may worsen under hormonal treatment or might interfere with the conduct of the study or the interpretation of the results (e.g., herpes gestationis or idiopathic icterus pregnancy; middle-ear deafness ; Sydenham's chorea, porphyria, disturbances in the bile flow.
* Liver diseases: Presence or history of severe hepatic diseases including benign or malignant tumors

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2006-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Bavaria, Germany

REFERENCES:
- [Result] Diefenbach K, Trummer D, Ebert F, Lissy M, Koch M, Rohde B, Blode H. EE-drospirenone-levomefolate calcium versus EE-drospirenone + folic acid: folate status during 24 weeks of treatment and over 20 weeks following treatment cessation. Int J Womens Health. 2013 Apr 11;5:149-63. doi: 10.2147/IJWH.S37254. Print 2013. PMID 23610531

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy female volunteers aged 18 - 40 (inclusive), desiring contraception, with Red Blood Cell folate > 317 nmol/L and < 906 nmol/L, with no concomitant intake of vitamin supplements or medication containing folate or interacting with folate, and no vitamin B12 deficiency, were enrolled from 11 December 2006 to 15 January 2008 at 1 German center
Pre-assignment Details: 235 female volunteers were screened according to the inclusion and exclusion criteria to determine that the volunteer was in a good state of health and appropriate for inclusion in the study, and 172 volunteers were randomized at one center.
Period: Overall Study
Arm/Group | EE 0.03 mg/DRSP 3 mg/Metafolin + Folic Acid Placebo | EE 0.03 mg/DRSP 3 mg (Yasmin) + Folic Acid
Started | 86 (randomized and received at least one dose of treatment) | 86 (randomized and received at least one dose of treatment)
Received Treatment | 79 | 82
Completed Treatment | 79 | 81
Completed | 75 (completed and valid for primary analysis data set) | 75 (completed and valid for primary analysis data set)
Not Completed | 11 | 11
Not completed — Adverse Event | 2 | 4
Not completed — Withdrawal by Subject | 3 | 0
Not completed — due to relocation | 2 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Invalid for primary analysis data set | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EE 0.03 mg/DRSP 3 mg/Metafolin + Folic Acid Placebo | EE 0.03 mg/DRSP 3 mg (Yasmin) + Folic Acid | Total
Number analyzed (Participants) | 86 | 86 | 172
Age Continuous [Mean (Standard Deviation); unit: years] | 28.4 (5.80) | 27.0 (5.49) | 27.7 (5.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 86 | 172
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) From Time 0 to 24 Weeks [AUC(0-24weeks)] for Plasma Folate and RBC (Red Blood Cell) Folate (Baseline Uncorrected)
Description: The Area under the curve (AUC) is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: up to 24 weeks of treatment
Measure: Geometric Mean (95% Confidence Interval); unit: nmol·week/L
Arm/Group | EE 0.03 mg/DRSP 3 mg/Metafolin + Folic Acid Placebo | EE 0.03 mg/DRSP 3 mg (Yasmin) + Folic Acid
Number analyzed (Participants) | 75 | 75
nmol·week/L
  plasma folate | 1030 [975 to 1087] | 904 [859 to 951]
  RBC folate | 24176 [23007 to 25405] | 21876 [21011 to 22776]

2. Primary Outcome: Area Under the Curve From Time 0 to 24 Weeks [AUC(0-24weeks)] for Plasma Folate and RBC (Red Blood Cell) Folate (Baseline Corrected)
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: up to 24 weeks of treatment
Measure: Geometric Mean (95% Confidence Interval); unit: nmol·week/L
Arm/Group | EE 0.03 mg/DRSP 3 mg/Metafolin + Folic Acid Placebo | EE 0.03 mg/DRSP 3 mg (Yasmin) + Folic Acid
Number analyzed (Participants) | 75 | 75
nmol·week/L
  plasma folate | 640 [600 to 684] | 561 [521 to 604]
  RBC folate | 10427 [9658 to 11258] | 8863 [8383 to 9370]

3. Primary Outcome: Proportion of Participants With RBC Folate Below 906 Nmol/L in the Yasmin + Metafolin Group in the Folate Elimination Phase (Week 24 to 44)
Description: Proportion of participants with RBC folate below 906 nmol/L in the Yasmin + Metafolin group in the folate elimination phase (week 24 to 44)
Time Frame: from week 24 to week 44
Measure: Number; unit: proportion of participants
Arm/Group | EE 0.03 mg/DRSP 3 mg/Metafolin + Folic Acid Placebo
Number analyzed (Participants) | 75
proportion of participants
  week 24 | 0.053
  week 26 | 0.067
  week 28 | 0.147
  week 30 | 0.213
  week 32 | 0.400
  week 34 | 0.533
  week 36 | 0.707
  week 38 | 0.760
  week 40 | 0.827
  week 42 | 0.867
  week 44 | 0.907

4. Secondary Outcome: Folate Metabolite Pattern in Plasma at Baseline
Description: Folate metabolite pattern in plasma at baseline
Time Frame: pre-treatment
Population: Note that not all samples were evaluable for each outcome measure. Therefore the number of participants analyzed not necessarily matches the number of completers.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | EE 0.03 mg/DRSP 3 mg/Metafolin + Folic Acid Placebo | EE 0.03 mg/DRSP 3 mg (Yasmin) + Folic Acid
Number analyzed (Participants) | 74 | 75
nmol/L
  Tetrahydrofolate (THF) | 4.07 (0.357) | 4.60 (0.656)
  5,10-methenyl-THF | 1.57 (0.412) | 1.63 (0.372)

5. Secondary Outcome: Folate Metabolite Pattern in Plasma at Cycle 3
Description: Folate metabolite pattern in plasma at cycle 3
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | EE 0.03 mg/DRSP 3 mg/Metafolin + Folic Acid Placebo | EE 0.03 mg/DRSP 3 mg (Yasmin) + Folic Acid
Number analyzed (Participants) | 75 | 75
nmol/L
  THF | 4.98 (1.851) | 5.28 (1.806)
  5,10-methenyl-THF | 1.76 (0.603) | 1.45 (0.282)

6. Secondary Outcome: Folate Metabolite Pattern in Plasma at Cycle 6
Description: Folate metabolite pattern in plasma at cycle 6
Time Frame: week 24
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | EE 0.03 mg/DRSP 3 mg/Metafolin + Folic Acid Placebo | EE 0.03 mg/DRSP 3 mg (Yasmin) + Folic Acid
Number analyzed (Participants) | 75 | 75
nmol/L
  THF | 5.92 (2.318) | 5.76 (2.835)
  5,10-methenyl-THF | 1.46 (0.238) | 1.95 (1.166)

7. Secondary Outcome: Homocysteine Concentrations in Plasma at Baseline and at the End of Treatment (Week 24) With Metafolin
Description: Homocysteine concentrations in plasma at baseline (median of baseline concentrations) and at the end of treatment (week 24) with Metafolin
Time Frame: baseline and week 24
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | EE 0.03 mg/DRSP 3 mg/Metafolin + Folic Acid Placebo
Number analyzed (Participants) | 75
µmol/L
  baseline | 9.3 (2.2)
  24 weeks | 7.5 (1.6)

8. Secondary Outcome: Homocysteine Concentrations in Plasma at Baseline and at the End of Treatment (Week 24) With Folic Acid
Description: Homocysteine concentrations in plasma at baseline (median of baseline concentrations) and at the end of treatment (week 24) with folic acid
Time Frame: baseline, and up to 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | EE 0.03 mg/DRSP 3 mg (Yasmin) + Folic Acid
Number analyzed (Participants) | 75
µmol/L
  baseline | 9.2 (1.9)
  24 weeks | 7.6 (1.4)

ADVERSE EVENTS:
Arm/Group | EE 0.03 mg/DRSP 3 mg/Metafolin + Folic Acid Placebo | EE 0.03 mg/DRSP 3 mg (Yasmin) + Folic Acid
Serious Adverse Events (participants affected / at risk) | 6/86 | 3/86
Other Adverse Events (participants affected / at risk) | 84/86 | 84/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EE 0.03 mg/DRSP 3 mg/Metafolin + Folic Acid Placebo (N=86) | EE 0.03 mg/DRSP 3 mg (Yasmin) + Folic Acid (N=86)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EE 0.03 mg/DRSP 3 mg/Metafolin + Folic Acid Placebo (N=86) | EE 0.03 mg/DRSP 3 mg (Yasmin) + Folic Acid (N=86)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 3 (3) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (3) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 4 (4)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Basedow's disease (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye allergy (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 6 (9)
Abdominal pain lower (Gastrointestinal disorders) | 1 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 5 (6)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 17 (21) | 19 (23)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Lip blister (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 14 (17) | 21 (27)
Oral mucosal blistering (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pruritus (Gastrointestinal disorders) | 1 (2) | 0 (0)
Radicular cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 8 (9) | 5 (6)
Vomiting (Gastrointestinal disorders) | 14 (14) | 17 (21)
Chills (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 7 (7)
Hunger (General disorders) | 1 (2) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (2) | 0 (0)
Puncture site pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 10 (10) | 6 (6)
Allergy to animal (Immune system disorders) | 2 (4) | 0 (0)
Seasonal allergy (Immune system disorders) | 7 (12) | 9 (13)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 1 (1) | 2 (2)
Anogenital warts (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (2)
Cystitis (Infections and infestations) | 4 (4) | 5 (7)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (6) | 8 (8)
Gastrointestinal infection (Infections and infestations) | 4 (4) | 6 (6)
Herpes dermatitis (Infections and infestations) | 1 (2) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 63 (106) | 60 (139)
Oral herpes (Infections and infestations) | 6 (7) | 9 (12)
Otitis media (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (2)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 8 (10) | 4 (5)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 3 (4) | 3 (3)
Tooth infection (Infections and infestations) | 2 (3) | 1 (1)
Vaginal candidiasis (Infections and infestations) | 4 (5) | 3 (3)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Ear canal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Whiplash injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 1 (2)
Electrocardiogram P wave abnormal (Investigations) | 0 (0) | 1 (1)
Serum ferritin decreased (Investigations) | 0 (0) | 2 (4)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (2) | 1 (1)
Food craving (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (10) | 5 (5)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 45 (122) | 53 (173)
Intercostal neuralgia (Nervous system disorders) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (2) | 0 (0)
Mood swings (Psychiatric disorders) | 2 (4) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 1 (2) | 0 (0)
Breast discomfort (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Breast disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast enlargement (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Breast pain (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Breast swelling (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 4 (6) | 7 (14)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menstruation delayed (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 6 (10) | 6 (7)
Nipple pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vulval disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (26) | 21 (26)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 (25) | 24 (35)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Photosensitivity allergic reaction (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Trichorrhexis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dental treatment (Surgical and medical procedures) | 3 (3) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Mole excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 1 (1) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 2 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI (principal investigator) of CRO (contract research organization) will refrain from publishing any data or information generated or derived as a result of the performance of the Services.